CLINICAL TRIAL: NCT03848793
Title: A Phase 2, Multiple Centers, Double-blind, Placebo-Controlled, Randomised Study to Evaluate the Efficacy and Safety of HS-20004 in Type 2 Diabetes Subjects.
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of HS-20004 in Type 2 Diabetes Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-20004-201
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-20004 or placebo treatment (Low dose) (Other): HS-20004 or placebo SC once daily (Low dose)
  Interventions: Drug: HS-20004
- HS-20004 or placebo treatment (median dose 1) (Other): HS-20004 or placebo SC once daily (median dose 1)
  Interventions: Drug: HS-20004
- HS-20004 or placebo treatment (median dose 2) (Other): HS-20004 or placebo SC once daily (median dose 2)
  Interventions: Drug: HS-20004
- HS-20004 or placebo treatment (high dose) (Other): HS-20004 or placebo SC once daily (high dose)
  Interventions: Drug: HS-20004

INTERVENTIONS:
Drug: HS-20004 — treatment
  Other Names: Noiiglutide Injection

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of Noiiglutide Injection as mono-therapy with different doses in subjects with type 2 diabetes compared to placebo for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed for more than 3 months
* HbA1c between 7.5 and 11.0 % (inclusive), and FPG ≥9.0mmol/l
* Body Mass Index (BMI) between 23 and 35 kg/m2(inclusive)

Exclusion Criteria：

* History or family history of drug allergy
* Subjects treated with any other anti-diabetes drug within 8 weeks before screening
* Participation in any other clinical trial of an investigational medicinal product within 3 months before screening
* Smoker or alcohol abuse
* Currently use or plan to use systemic corticosteroid
* History of recurrent severe hypoglycemia
* Type 1 diabetes or secondary diabetes mellitus
* Uncontrolled active or untreated hypertension
* History of pancreatitis (acute or chronic)
* Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN2) or Medullary Thyroid Carcinoma (MTC)
* Serious unconscious hypoglycemia history
* Within the past 6 months before screening any of the following: coronary artery revascularization, patients presently classified as being in New York Heart Association (NYHA) Class III or IV, myocardial infarction, stroke or unstable angina and/or persistent and clinically significant arrhythmias
* Female subject of childbearing potential who does not use an acceptable method of birth control, is pregnant or planning a pregnancy, or breastfeeding, or male subject who does not use an acceptable method of birth control
* Subject was not used for the study as determined by the Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks treatment
  Estimated mean change from baseline in HbA1c at week 16. The data were analysed for the "on-treatment until rescue medication" observation period which includes observations recorded at or after date of first dose of trial product

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose | 16 weeks treatment
  Estimated mean change from baseline in FPG at week 16.
Change in Body Weight | 16 weeks treatment
  Estimated mean change from baseline in Body Weigh at week 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No